CLINICAL TRIAL: NCT04514536
Title: Combinatorial Approach of Connected Functions for Multimodal Health Data Collection
Brief Title: Evaluation of a Health Monitoring Platform for Elderly in Home Care Context
Acronym: ACCORDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Collaborators: AZNetwork (Unknown); RF-Track (Unknown); LTSI Rennes (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A02316-51
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Aging; Frailty
Keywords: Health monitoring; Frailty; Home care; Home support
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health monitoring (Experimental): Subjects have to monitor their health autonomously using the monitoring platform (connected health devices and app on the touchpad).
  Interventions: Device: Health monitors

INTERVENTIONS:
Device: Health monitors — * The connected scale (iHealth HS2) measures weight from 5 to 180kg and BMI.
  * The connected actimeter (iHealth AM4) monitors activity (number of steps, distance, calories), sleep (automatic sleep recognition, effective sleep time, number of awakenings) and swimming (automatic activity recognition, session duration, swim type recognition and number of laps).
  * The connected blood pressure monitor (iHealth Track KN-550BT)is a medical device that measures blood pressure and pulse rate.
  * The activity monitor (manufactured by RF Track) consists of a housing that can be positioned as a pendant or at the hip. It includes an accelerometer, gyroscope, magnetometer, barometer, radio transceiver, and led. The sensor records the raw signals.
  * The touchpad allows the subject to connect to the Calliope app. This app allows the data recovery, storage, analysis, visualization, and all the required settings for the platform to work together.

SUMMARY:
This study aims at, as a primary objective, studying acceptability of elderly about a health monitoring platform for home support and home care. The secondary objective consists in studying the correlation of different health data evolution and the frailty trajectory of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years old
* Living at home or in senior residence
* Evaluated as being robust according to the Fried's frailty test (0 met criteria)
* Affiliated or beneficiary of a social protection scheme
* Having given written consent

Exclusion Criteria:

* Hospitalization during the month preceding the first visit
* Subject suffering from cognitive disorders preventing proper use of the device
* Subject being unable to give by himself / herself his / her consent to participate in the trial
* Person subject to legal protection (safeguard of justice, trusteeship, guardianship, persons deprived of liberty)

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Beliefs modified questionnaire | 1 month
  questionnaire by Fishbein & Ajzen (1975), is a qualitative questionnaire, with no scoring
UTAUT modified questionnaire | 1 month
  questionnaire by Venkatesh et al. (2003) Final score is graded 1 to 10, 10 being the best score
Usability SUS questionnaire | 1 month
  questionnaire by Brooks (1996) Final score is graded 10 to 70, 70 being the best score
Comfort modified questionnaire | 1 month
  questionnaire by Knight & Baber (2005) Final score is graded 11 to 77, 77 being the best score

SECONDARY OUTCOMES:
Motivation modified questionnaire | inclusion
  questionnaire by Deci & Ryan (1987), is a qualitative questionnaire, with no scoring
Beliefs modified questionnaire | inclusion
  questionnaire by Fishbein & Ajzen (1975), is a qualitative questionnaire, with no scoring
Beliefs modified questionnaire | 12 months
  a priori acceptability questionnaire by Fishbein & Ajzen (1975), is a qualitative questionnaire, with no scoring
Beliefs modified questionnaire | 24 months
  a priori acceptability questionnaire by Fishbein & Ajzen (1975), is a qualitative questionnaire, with no scoring
UTAUT modified questionnaire | inclusion
  questionnaire by Venkatesh et al. (2003) Final score is graded 1 to 10, 10 being the best score
UTAUT modified questionnaire | 12 months
  questionnaire by Venkatesh et al. (2003) Final score is graded 1 to 10, 10 being the best score
UTAUT modified questionnaire | 24 months
  questionnaire by Venkatesh et al. (2003) Final score is graded 1 to 10, 10 being the best score
Comfort modified questionnaire | inclusion
  questionnaire by Knight & Baber (2005) Final score is graded 11 to 77, 77 being the best score
Comfort modified questionnaire | 12 months
  questionnaire by Knight & Baber (2005) Final score is graded 11 to 77, 77 being the best score
Comfort modified questionnaire | 24 months
  questionnaire by Knight & Baber (2005) Final score is graded 11 to 77, 77 being the best score
Usability SUS questionnaire | inclusion
  questionnaire by Brooks (1996) Final score is graded 10 to 70, 70 being the best score
Usability SUS questionnaire | 12 months
  questionnaire by Brooks (1996) Final score is graded 10 to 70, 70 being the best score
Usability SUS questionnaire | 24 months
  questionnaire by Brooks (1996) Final score is graded 10 to 70, 70 being the best score

CONTACTS AND LOCATIONS:
Overall Officials: Dominique SOMME, MD, PhD, Principal Investigator — Rennes University Hospital